CLINICAL TRIAL: NCT04550793
Title: Using Shear Wave Ultrasound Elastography for Follow up After Anti-spastic Intervention Among Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202006138RINB
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-07

CONDITIONS: Stroke; Spasticity, Muscle; Botulism; Ultrasound; Activity of Daily Living
MeSH Terms: conditions — Stroke; Muscle Spasticity; Botulism | interventions — Botulinum Toxins

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention: The stroke patients who receive botulinum toxin injection at affected brachialis and/or biceps brachials.
  Interventions: Drug: Botulinum toxin injection
- Control: The stroke patients who do not receive botulinum toxin injection at affected brachialis and/or biceps brachials in the past 3 months.

INTERVENTIONS:
Drug: Botulinum toxin injection — Botulinum toxin injection at affected brachialis and/or biceps brachials.
  Groups: Intervention

SUMMARY:
Spasticity of stroke patient, a very common complication in clinical practice, affects performance of hand function and gait pattern. It also interferes with quality of life of patients severely. Currently first line clinical approach to spasticity consist of physical therapy and pharmacological management. However, there are still some refractory cases that needed local intervention such as Botox injection.

So far, we only can use subjective methods to measure muscle tension, such as modified Ashworth scale and Tone Assessment Scale. In our previous study, we found that ultrasound shear wave image could correlate with muscle stiffness caused by poststroke spasticity. With this new method, we aim to establish a more objective method in measuring abnormal poststroke muscle tension before and after treatments and further monitor therapeutic effect. We also include several assessment scales to evaluate the correlation between measured muscle spasm and activity of daily living.

We hypothesize that the rheological changes in muscles muscle spasm after Botox injection can be detected by ultrasound shear wave image. Therapeutic effect can also be seen in its effect on daily functions.

In this project, we will use shear wave imaging of ultrasound to investigate the elasticity (and hardness) of the biceps brachii and brachialis muscle in stroke patients with unilateral hemiplegia before and after Botox injection. The findings of this project will provide the objective evaluation of muscle spasticity and its correlation with functional status, which will provide new points of view toward treatment of spasticity.

ELIGIBILITY:
Inclusion Criteria:

[Intervention group]

* Stroke patients with unilateral involvement
* Patient's spasticity over affected upper extremities scored at least 1+ with Modified Ashworth Scale
* Patient required botulinum toxin injection at affected upper limb muscle per primary care physician.

[Control group]

* Stroke patients with unilateral involvement
* Patient's spasticity over affected upper extremities scored at least 1+ with Modified Ashworth Scale

Exclusion Criteria:

* Patients ever diagnosed with cerebral diseases other than stroke, such as traumatic brain injury, encephalitis and brain tumor
* Patients failed to cooperated due to cognition, consciousness or speech problem
* Patients with illness that could affect muscle stiffness, such as spinal cord injury and Parkinson's disease
* Patients with upper limb contracture
* Patients receiving botulinum toxin injection or shock wave therapy over upper extremities during past three months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patient aged above 20 years old with unilateral involvement.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Shear Wave Ultrasound Elastography | During each follow up visit within 12 weeks time frame
  Shear wave ultrasound elastography measurement of spastic upper limb muscles, including biceps brachii and brachialis

SECONDARY OUTCOMES:
Barthel Index (Wade's version) | During each follow up visit within 12 weeks time frame
  Barthel Index assessing activities of daily livings
Revised Nottingham Extended Activities of Daily Livings Scale | During each follow up visit within 12 weeks time frame
  Revised Nottingham Extended Scale assessing activities of daily livings
Stroke Rehabilitation Assessment of Movement (STREAM), brief version | During each follow up visit within 12 weeks time frame
  STREAM assessing movement condition
Modified Ashworth Scale (MAS) | During each follow up visit within 12 weeks time frame
  MAS scale for assessing spasticity
Tone Assessment Scale (TAS) | During each follow up visit within 12 weeks time frame
  TAS scale for assessing spasticity
Global improvement scale | During each follow up visit within 12 weeks time frame
  Global improvement scale for assessing symptoms related to stroke
Self-report spasticity symptoms | During each follow up visit within 12 weeks time frame
  Self-report spasticity symptoms for assessing spasticity
EuroQol | During each follow up visit within 12 weeks time frame
  EuroQol for evaluating quality of life
Extended Activities of Daily Living | During each follow up visit within 12 weeks time frame
  Extended Activities of Daily Living scale for evaluating activity of daily living
Postural Assessment Scale for Stroke Patients (PASS), brief version | During each follow up visit within 12 weeks time frame
  PASS for evaluating symptoms related to stroke

CONTACTS AND LOCATIONS:
Overall Officials: Huey-Wen Liang, MD PHD, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No